CLINICAL TRIAL: NCT05942716
Title: Involvement of the Serotonergic System in the Control of Impulsivity in Tourette Disorder.
Brief Title: Serotonin Control of Impulsivity in Tourette Disorder
Acronym: ARITEP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL22_0683
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Tourette Disorder
Keywords: Tourette; Serotonin; Impulsivity; Neuroimaging
MeSH Terms: conditions — Tourette Syndrome; Impulsive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tourette disorder (Experimental): 25 mixt adult patients with TD. Patients will be recruited if a current treatment by aripiprazole (5-15 mg) is already scheduled before the study.
  Interventions: Drug: Administration of a PET radiotracer

INTERVENTIONS:
Drug: Administration of a PET radiotracer — A highly selective 5-HT2A receptor ligand ([18F]-altanserin) will be injected to patients before each PET scan. The IV injection in the arm (via a catheter) will be performed in continue during a period of 2 hours in the imaging centre (CERMEP) before the acquisition. The dose will be 2,6 MBq/kg +/- 10 % depending the prescription of the nuclear medicine.
  Patients will be evaluated twice, one time free of neuroleptic treatment and a second time during stable chronic treatment by neuroleptic.

SUMMARY:
Tourette disorder (TD) is a neurodevelopmental disorder characterized by motor and vocal tics. It is often associated with multiple psychiatric comorbidities involving a high degree of impulsivity such as obsessive-compulsive disorders (OCD), attention-deficit hyperactivity disorders (ADHD), and intermittent explosive disorders (IED). Although a substantial body of clinical studies have emphasized the role of the dopamine system in motor symptoms, little is known about how the serotonergic (5-HT) system modulate both cognitive and affective abilities in TD. Several lines of evidence suggest that different 5-HT receptor subtypes may constitute a crucial factor in the development and maintenance of different symptoms. Because abnormal 5-HT2A receptor bindings have been reported in patients with TD and aripiprazole (drug of first choice) is a 5-HT2A antagonist, we hypothesize that 5-HT2A receptors may play an important role in regulating psychiatric symptoms in TD such as those characterized by impulsive behaviors. To investigate the involvement of 5-HT2A receptors in TD, we propose to perform a multimodal imaging study with 20 adult patients (ON and OFF treatment). Neuroimaging data will be collected with a hybrid system that simultaneously combines the positron emission tomography (PET) and the functional magnetic resonance imaging (fMRI). A highly selective PET radiotracer ([18F]-altanserin) will map 5-HT2A receptor bindings in the whole brain, while fMRI will provide detail information regarding the altered brain activities.

ELIGIBILITY:
* Inclusion Criteria * :

  * Male or Female
  * Diagnosed with a Tourette Disorder following the DSM-5
  * Age between 18-65 years
  * Member of a social security scheme in France
  * Freely-given informed consent to participate to this study (written form)
  * With a current treatment by aripiprazole already scheduled
  * With Tics compatible with TEP/fMRI exams
  * Having (for women only) effective contraception throughout participation in the study.

Exclusion Criteria * :

* Male or Female
* A serious not controlled psychiatric comorbidity
* A serious, evolving or debilitating pathology with a potential influence on the study
* Drug-taking with serotonergic effects (e.g., amphetamine, cocaine, MDMA, SSRIs, mianserin)
* Contraindication for fMRI and PET (e.g., pacemaker, ferromagnetic implant, claustrophobia)
* Women breastfeeding
* Protected or restricted person (administratively or in judicial terms)
* Participants to another study with radiations or radiotracers since less of one year, participants to a concomitant study
* Do not speak french

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2027-09-24 (Estimated); Study Completion 2028-09-24 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficients between receptor-specific imaging data (PET) and scores of impulsivity measured by the Barratt scale (BIS11). | As the analysis requires a complex imaging processing, this outcome measure will be assessed in the year following the acquisition.
  Correlation coefficients between changes in the binding potential (BPND) of [18F]-altanserin measured voxel-by-voxel in the whole brain and the evolution of scores BIS11 in TD patients.

SECONDARY OUTCOMES:
Correlation coefficients between receptor-specific imaging data (PET) and other clinical/behavioral scores. | As the analysis requires a complex imaging processing, this outcome measure will be assessed in the year following the acquisition.
  Correlation coefficients between changes in the binding potential (BPND) of [18F]-altanserin measured voxel-by-voxel in the whole brain and the evolution of other clinical scores and task performance of TD patients.
Correlation coefficients between functional imaging data (fMRI) and scores of impulsivity measured by the Barratt scale (BIS11). | As the analysis requires a complex imaging processing, this outcome measure will be assessed in the year following the acquisition.
  Correlation coefficients between changes in the BOLD signal measured voxel-by-voxel in the whole brain and the evolution of scores BIS11 in TD patients.
Correlation coefficients between functional imaging data (fMRI) and other clinical/behavioral scores. | As the analysis requires a complex imaging processing, this outcome measure will be assessed in the year following the acquisition.
  Correlation coefficients between changes in the BOLD signal measured voxel-by-voxel in the whole brain and the evolution of other clinical scores and task performance of TD patients.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service de neurologie C Hôpital neurologique Pierre Wertheimer/GHE Hospices Civils de Lyon, Bron
  - Centre de Référence Syndrome Gilles de la Tourette Département de Neurologie Pôle des Maladies du Système Nerveux Hôpital de la Pitié-Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: Undecided